CLINICAL TRIAL: NCT04430985
Title: FOLFOX + Immunotherapy With Intrahepatic Administration of Oxaliplatin for Patients With Multiple Non-resectable Liver Metastasis From Colorectal Cancer
Brief Title: FOLFOX + Immunotherapy With Intrahepatic Oxaliplatin for Patients With Metastatic Colorectal Cancer
Acronym: IMMUNOX
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Problems identifying eligble patients
Sponsor: Dorte Nielsen (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Dorte Nielsen, Professor Dorte Nielsen, MD, PhD, DMSc, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI 1949; 2019-004397-26 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOX + Immunotherapy (Experimental): 8 cycles of FOLFOX every 2 weeks with intrahepatic administration of oxaliplatin in cycles 1-4, thereafter (cycles 5-8) oxaliplatin i given i.v.; starting from cycle 3 this is combined with i.v. administration of nivolumab (cycle 3-8) and ipilimumab (cycle 3 + 6)
  Immunotherapy:
  Starting from cycle 3: Nivolumab 3 mg/kg i.v. on day 3 (every 2nd week, total of 6 administrations), Ipilimumab 1 mg/kg i.v. on day 3 (every 6th week, total of 2 administrations)
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Nivolumab; Device: Ipilimumab

INTERVENTIONS:
Drug: Oxaliplatin — Day 1 in cycle 1-4: 100 mg/m2 intrahepatic administration Day 1 in cycle 5-8: oxaliplatin 85 mg/m2 i.v.
Drug: 5-Fluorouracil — Day 1 each cycle: 400 mg/m2 i.v. bolus, 2400 mg/m2 i.v.over 46 hrs
Drug: Leucovorin — Day 1 each cycle: 400 mg/m2 i.v.
Drug: Nivolumab — Day 3 in cycle 3 to 8: 3 mg/kg i.v.
Device: Ipilimumab — Day 3 in cycle 3 and 6: 1 mg/kg i.v.

SUMMARY:
In this trial chemotherapy regimen FOLFOX with intrahepatic administration of oxaliplatin is combined with immunotherapy (nivolumab and ipilimumab) for the group of patients with multiple liver metastasis from colorectal cancer. Investigators hope to increase the disease-free survival after 3 years from 10 % to 30%.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age: 18 - 79 years
* Performance status 0-1.
* Histologically documented colorectal cancer (In case primary tumor has not yet been removed, it should be possible to be removed by surgery)
* Tumor is immunohistochemically microsatellite stable (MSS)
* More than 5 liver metastasis, not eligible for liver resection or radiofrequency ablation (RFA)
* Presence of liver metastasis documented on CT-scan with no documented extrahepatic disease except from primary tumor in situ.
* Measurable disease according to RECIST 1.1
* Involved liver tissue under 70 %
* Perfusion of liver metastasis possible via a. hepatica
* ANC >= 1,5 x 10¨9/ml og Platelets >= 100 x 10¨9/ml ,
* Estimated creatinine clearance >= 60 ml/min
* INR < 1,4 and bilirubin <= 1,5 x ULN

Exclusion Criteria:

* Current or prior second malignancy within 5 years, except from basal cell carcinoma or carcinoma in situ cervix uteri.
* Severe medical condition, such as severe cardiac disease or AMI within 1 year
* Uncontrolled infection.
* Patients positive for HIV, HBV-sAG or HCV antibody
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of ipilimumab, nivolumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, or topical steroids; or local steroid injections (e.g. intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Patients requiring treatment with oral prednisolon of dose > 10 mg daily
* Previous severe, unexpected reaction related to treatment with fluoropyrimidine.
* Previous treatment with oxaliplatin or immunotherapy
* Neuropathy that is contraindicated for treatment with oxaliplatin
* Pregnant or breastfeeding women. Women with childbearing potential (WOCBP) should have a negative pregnancy test and agree to use highly effective method(s) of contraception during treatment and 6 months thereafter.
* Men who are sexually active with WOCBP who do not agree to use highly effective method(s) of contraception during treatment and 7 months after immunotherapy or 6 months after chemotherapy (which period is the longest)
* Patients who, for linguistic, intellectual or cultural reasons, will not be able to fully understand the concept of treatment and respond to any. complications.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Disease-free Survival at 3 years | 3 years from start of treatment within the trial
  Proportion of patients without signs of disease 3 years after treatment start

SECONDARY OUTCOMES:
Patients becoming eligible for resection of liver metastasis | Evaluation of resectability after 8 cycles (each cycle is 14 days) of treatment (i.e after 16 weeks)
  Number of patients with reduction of tumor burden to an extent that they become eligible for resection/radio frequency ablation of liver metastasis
Objective response rate | Evaluation by CT-scan after 8 cycles (each cycle is 14 days) of treatment (i.e after 16 weeks)
  Proportion of patients with complete or partial response according to RECIST v1.1
Progression free survival | Evaluation by CT-scan after 8 cycles of treatment each cycle is 14 days) and every 3 months thereafter until progression (max 3 years)
  Time from start of treatment to progression of disease or death
Overall survival | Survival follow-up is planned for at least 3 years from treatment start
  Time from start of treatment to death
Safety and tolerability of the treatment | During the 16 weeks of treatment and 100 days thereafter (up to 31 weeks)
  Incidence of treatment related Adverse Events

OTHER OUTCOMES:
Exploratory analysis of immunological response in tumor tissue | Tumor tissue samples taken at baseline and week 16
  Composition of immune infiltrates in order to define the immune cell subsets present within FFPE tumor tissue before and after exposure to therapy.
Explorative analysis of biomarkers predictive of response to the combination of nivolumab, ipilimumab in combination with FOLFOX | Blood samples are drawn at baseline through study completion (up to 3 years)
  Biomarker analyses include, but are not limited to a range of molecules with different characteristics such as DNA, Single Nucleotide Polymorphism (SNPs), RNA, microRNA, proteins and metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Ole Larsen, MD, PhD, Principal Investigator — Herlev Hospital, Department of Oncology
Locations (1):
- Herlev University Hospital, Department of Oncology, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No